CLINICAL TRIAL: NCT06399276
Title: A Proof-of-Concept Study Evaluating a 4:3 Intermittent Fasting Weight Loss Intervention in Adults With Breast Cancer and Overweight or Obesity
Brief Title: 4:3 Intermittent Fasting Intervention in Adults With Breast Cancer and Overweight or Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-1546.cc; R01CA258766 (NIH)
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Overweight; Obese
MeSH Terms: conditions — Breast Neoplasms; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Weight Loss Focused on Intermittent Fasting (Experimental): 3-month integrated behavioral weight loss intervention with a dietary focus on intermittent fasting.
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Behavioral: Weight Loss — Participants are instructed to perform a modified fast (~500 kcal) on 3 days/week with ad libitum intake the other 4 days/week. Group-based behavioral support sessions will be held by an experienced Registered Dietician. Participants will attend BfitBwell exercise sessions in person and virtually to receive individualized support to progress to 150 min/wk of moderate-intensity physical activity

SUMMARY:
This is a 3 month single arm pilot and feasibility study designed to examine the impact of an intermittent fasting lifestyle weight loss intervention on pre-specified clinical milestones (change in body weight, adherence to the fasting program, and moderate-to vigorous physical activity, MVPA) in adults with overweight and obesity and breast cancer after they have completed their cancer treatment. The investigators will also evaluate feasibility of recruitment and retention of study participants, safety of the intervention, and obtain feedback from participants to improve the program. Participants will receive a 3 month lifestyle weight loss program focusing on a 4:3 intermittent fasting paradigm (3 modified fast days per week) and support to increase physical activity to 150 minutes per week. Outcome measures will be assessed at the end of the 3 month intervention (primary endpoint) and after a 3 month weight maintenance follow up phase.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Age 18-65 years
* Body Mass Index 25-45 kg/m2
* Diagnosis of stage 1-3 breast cancer within the past 10 years with completion of standard of care definitive surgery, adjuvant chemotherapy, radiation, immunotherapy and/or targeted therapy as appropriate prior to the intervention start date. Completion of definitive surgery must be ≥ 3 months prior to the intervention start date, other therapies must be completed ≥ 1 month prior to the intervention start date (however exceptions to this 1-month timeframe for completion of other therapies can be made on a case-by-case basis by the PI if patients are tolerating therapy without adverse effects and will have completed treatment prior to the intervention start date). Current/ongoing use of anti-endocrine directed therapy for breast cancer (including ovarian suppression, tamoxifen, aromatase inhibitors, selective estrogen degraders) is acceptable as long as participants have been on therapy for ≥3 months prior to the intervention start date.
* Live or work within 30 miles of the AHWC (exceptions may be made at the discretion of the Study PI on a case-by-case basis for highly motivated subjects).
* Capable and willing to give informed consent and understand exclusion criteria, willing to attend weekly small group sessions held by a registered dietitian, and attend one in person BfitBwell exercise sessions per week.
* Have a primary care provider (PCP) (or are willing to establish care with a PCP prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions.
* Obtain a signed medical clearance from their medical provider for participation in the 4:3 IMF dietary intervention and BfitBwell clinical exercise oncology program.
* Own or willing to purchase a smart phone or computer to join Zoom meetings, complete questionnaires, and access/download the True Coach virtual exercise coaching sessions.

All interested individuals will complete a brief online eligibility screener through REDCap to confirm initial eligibility.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 2 or higher.
* Actively undergoing chemotherapy, radiation, immunotherapy and/or targeted therapy (other than anti-endocrine therapy) or are within 1 month of completion of chemotherapy, radiation, immunotherapy and/or targeted therapy (other than anti-endocrine therapy) as of the target intervention start date. Exceptions to this 1-month timeframe can be made on a case-by-case basis at the discretion of the PI if patients are tolerating therapy without adverse effects and will have completed treatment prior to the intervention start date.
* Plans to relocate within the next 12 months.
* Plans for extended travel (>2 weeks) within the next 12 months.
* Major surgery within the past 3 months (including mastectomy or breast reconstruction but not including lumpectomy or other minor surgeries) or planned major surgery (including mastectomy or breast reconstruction) during the timeframe of the 6 month study intervention and follow-up phases.
* For Females:

  * Currently pregnant or lactating.
  * Pregnant within the past 6 months.
  * Planning to become pregnant in the next 12 months; sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception.
* Recent (past 6 months) acute coronary event, unstable angina, coronary revascularization, stroke, pulmonary embolism, or hospitalization for heart failure or cardiac arrythmia.
* Symptoms suggestive of cardiovascular disease or unstable angina (e.g., chest pain, shortness of breath at rest or with mild exertion, lightheadedness, syncope).
* Uncontrolled hypertension, defined as diastolic blood pressure >100 mmHG, systolic blood pressure >160 mmHG, or resting heart rate >100 bpm as measured in duplicate on the screening visit after 5 minutes of rest in a seated position.
* Diabetes (history of type 1 or type 2 diabetes or fasting glucose ≥126 mg/dL or Hemoglobin A1C ≥6.5% as measured on screening labs) unless on metformin or on dipeptidyl peptidase IV (DPP-IV) inhibitor monotherapy and well-controlled with Hemoglobin A1C <8%.
* Undiagnosed hypo- or hyper-thyroidism (TSH outside of the normal range as measured on screening labs) or history of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen is acceptable.
* Stage 4 or 5 chronic kidney disease as assessed by estimated glomerular filtration rate <30 as measured on screening labs.
* Triglycerides >500 mg/dL or LDL cholesterol >200 mg/dL as measured on screening labs.
* Serious arrhythmias, including multifocal PVC's, frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, known QTc interval > 480 msec or other significant conduction defects.
* Clinically significant abnormalities in hematocrit/hemoglobin, white blood cell count, platelets, serum sodium, potassium, or bicarbonate as measured on screening labs or presence or history of other metabolic or chronic health problems which would impact ability to safely participate in a weight loss intervention involving an intermittent energy restricted diet and exercise including significant cardiac valvular disease or heart failure, significant gastrointestinal, pulmonary, renal, musculoskeletal, neurologic, hematologic, orthopedic, or psychiatric disease.
* Sustained use of prescription or over-the-counter medications known to significantly impact appetite, weight, or energy metabolism (e.g., anti-obesity pharmacotherapy, appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants) with the exception of anti-endocrine directed treatment for breast cancer and standard of care anti-emetic or anti-diarrheal agents.
* Sustained use of systemic glucocorticoids (current or in the past 6 months) unless physiologic replacement therapy for adrenal insufficiency.
* Previous obesity treatment with metabolic bariatric surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.
* Nicotine use (current or past 6 months)
* Current alcohol or substance abuse.
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the Eating Attitudes Test (EATS-26) or pattern of response on the Questionnaire of Eating and Weight Patterns (QEWP-5) suggestive of possible binge eating disorder or bulimia will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode or history of other significant psychiatric illness (e.g., psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study PI would interfere with ability to participate in the diet and exercise interventions and provide feedback on the interventions via questionnaires and focus groups.
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials over the next 12 months.
* Previous participation (within the past 3 years) in the Anschutz Health and Wellness Center (AHWC) BfitBwell Oncology Exercise Program (exceptions may be made at the discretion of the study PI).
* Previous participation (within the past 3 years) in a weight loss, exercise, or nutrition research study (exceptions may be made at the discretion of the study PI).

Children (individuals under the age of 18 years per NIH guidelines) will not be recruited for the current studies because breast cancer is rare in children and because the lifestyle weight management curriculum used in the study was not designed for children or adolescents.

We have elected to exclude adults over the age of 65 years as weight loss may not be advisable in older patients undergoing treatment for breast cancer or in routine follow-up for breast cancer due to issues with loss of lean mass and decreases in functional capacity that can occur with weight loss in older individuals. A separate study on the impact of a lifestyle weight loss intervention in older patients with breast cancer is warranted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 3 months
  Measured using digital scale accurate to =/-0.1 kg, in the morning in a fasted state
Adherence to 4:3 Intermittent Fasting Dietary Paradigm as Measured by Food Records | 3 months
  Dietary energy intake assessed using written food records for 7 consecutive days
Physical Activity | 3 months
  Moderate to Vigorous Physical Activity (MVPA) (min/wk) measured with the activPALv4 activity monitor for 7 consecutive days.

SECONDARY OUTCOMES:
Rate of Enrollment | at recruitment
  Number of participants enrolled per month during the recruitment phase.
Percent of Participants Completing Outcome Measures | 3 months
  Retention of participants in the 3-month intervention assessed by percent of enrolled participants that complete outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Catenacci, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Anschutz Health and Wellness, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado